CLINICAL TRIAL: NCT03685526
Title: Evaluation of the Cinenses Lung Volume Reduction Reverser System in Treating Patients With Severe Emphysema
Brief Title: Cinenses Lung Volume Reduction Reverser System First-in-man Study Treating Patients With Severe Emphysema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LVR-EU-FIM-01
Record Dates: First submitted 2018-09-17; First posted 2018-09-26 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Patients will be treated with Cinenses Lung Volume Reduction Reverser System.
  Interventions: Device: Cinenses Lung Volume Reduction Reverser System

INTERVENTIONS:
Device: Cinenses Lung Volume Reduction Reverser System — Lung Volume Reduction Reverser System is show as figure 1-4, consists of lung volume reduction reverser (short as: reverser), conveyor, measuring guide wire and transporting sheath. Matrix of reverser is nickel titanium alloy, its surface is coated by polymer flexible film, at the end of the connection segment is specially designed connector, which is easy for the reverser's transport and recycling. The silica gel part at the far end of reverser makes it softer.

SUMMARY:
The study is designed as a prospective, nonrandomized, exploratory, single center, first-in-man study. The objective of this study is to evaluate its safety and feasibility of the CinensesTM Lung Volume Reduction Reverser System in patients with severe emphysema. The study will also collect clinical data up to 6-month follow-up to explore its safety and effectiveness.

DETAILED DESCRIPTION:
The study is designed as a prospective, nonrandomized, exploratory, single center, first-in-man study. The objective of this study is to evaluate its safety and feasibility of the CinensesTM Lung Volume Reduction Reverser System in patients with severe emphysema. The study will also collect clinical data up to 6-month follow-up to explore its safety and effectiveness. Study Population ：Patients with severe emphysema and have to meet all the inclusion and exclusion criteria.

Sample Size： 15 subjects

ELIGIBILITY:
Candidates for this study must meet all of the following inclusion criteria:

1. Patient between 50 to 80 years old
2. High Resolution CT scan indicates homogeneous or heterogeneous emphysema.
3. Patient has post- bronchodilator FEV1 less than or equal to 45% of predicted
4. Total Lung Capacity > 100% of predicted.
5. Residual volume≥ 200% of predicted.
6. Patient has marked dyspnea scoring >2 on mMRC scale of 0-4.
7. Patient has stopped smoking for a minimum of 8 weeks prior to entering the study, as confirmed by COHb ≤2.5%
8. Patient (and legal guardian if applicable) read, understood and signed the Informed Consent form.
9. Subject has completed a pulmonary rehab within the last year and/or performs regularly physical activity.

Candidates will be excluded from the study if any of the following conditions are present:

1. Patient has a change in FEV1 > 20% post-bronchodilator
2. Patient has a history of recurrent clinically significant respiratory infection, defined as with more than 3 hospital stays in the past 12 months.
3. Patient has uncontrolled pulmonary hypertension defined by right ventricular pressure>50mmHg and/or evidenced by echocardiogram.
4. Patient has an inability to walk >140 meters (150 yards) in 6 minutes.
5. Patient has evidence of any other disease that may compromise survival such as lung cancer, renal failure, any other investigator identified such evidences.
6. Patient is pregnant or lactating.
7. Patient has an inability to tolerate bronchoscopy under anesthesia.
8. Any contraindication to bronchoscopy procedure, including but not limited to:

   1. Untreatable life-threatening arrhythmias
   2. Inability to adequately oxygenate the patient during the procedure
   3. Acute respiratory failure with hypercapnia
   4. Within 6 months myocardial infarction
   5. Previously diagnosed high-grade tracheal obstruction
   6. Uncorrectable coagulopathy
9. Patient has clinically significant bronchiectasis.
10. Patient has giant bullae > 1/3 lung volume.
11. Patient has had previous LVR surgery, lung transplant or lobectomy，or has still ELVR devices or other device to treat COPD in either lung.
12. Patient has been involved in other clinical studies within 30 days prior to this study.
13. Patient is taking > 20mg prednisone (or similar steroid) daily.
14. Patient on antiplatelet agent (eg, clopidogrel) or anticoagulant therapy (eg, heparin or coumadin) or has not been weaned off prior to procedure.
15. Patient has any other disease that would interfere with completion of study, follow up assessments or that would adversely affect outcomes.
16. A known allergy to nitinol.
17. Patient with uncontrolled diabetes as well as overweight patient (BMI > 35 kg/m2)
18. Cancer needs chemotherapy in past two years
19. Patient with pleural effusion and/or pneumothorax
20. Patient with a disease history of asthma, cystic fibrosis, interstitial lung disease (ILD), active tuberculosis;
21. Patient with exacerbation of chronic obstructive pulmonary disease (COPD) which defined as: An acute event with the need of antibiotic treatment or hospitalization.
22. Subject has severe gas exchange abnormalities as defined by:

    PaCO2 >55 mm Hg,PaO2 <45 mm Hg on room air
23. Patient with acute ischemic heart disease, with proven pulmonary hypertension (SPAP> 45 mmHg) in echocardiography and/or need for double platelet aggregation inhibition

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient between 50 to 80 years old
Enrollment: 15 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 3-month post final bronchoscopy
  Evaluate adverse events associated with implantation of the Cinenses Lung Volume Reduction Reverser System at 3-month post final bronchoscopy. CinensesTMLung Volume Reduction Reverser System at 3-month post final bronchoscopy.

SECONDARY OUTCOMES:
Device success (Device level) | immediate postoperative
  Device success was defined as successful delivery and deployment of the study device at the intended target position and successful withdrawal of the delivery system.
Procedural success | during the hospital stay
  Procedural success was defined as all the study devices that were intended to be used during one procedure were achieved device success and the subject was without the occurrence of device-related or procedure-related SAEs during the hospital stay
St. George's Respiratory Questionnaire (SGRQ) score | 1,3,6-month,12-month follow-up
  The improvement of St. George's Respiratory Questionnaire (SGRQ) score from baseline (Pre-Treatment Visit) to 1-, 3- and 6-month ,12-month follow-up.
Percent change in forced expiratory volume in 1 second | 1,3,6-month,12-month follow-up
  Percent change in forced expiratory volume in 1 second (FEV1) from baseline (Pre- Treatment Visit) compared to 1-, 3- and 6-month,12-month follow-up.
Decrease in the Residual Volume (RV) | 1,3,6-month,12-month follow-up
  Decrease in the Residual Volume (RV) from baseline (Pre-Treatment Visit) compared to
  1-, 3- and 6-month,12-month follow-up.
Improvement in the 6-minute walk test | 1,3,6-month,12-month follow-up
  Improvement in the 6-minute walk test from baseline (Pre-Treatment Visit) compared to
  1-, 3- and 6-month,12-month follow-up
Improvement in the mMRC dyspnea scale | 1,3,6-month,12-month follow-up
  Improvement in the mMRC dyspnea scale from baseline (Pre-Treatment Visit) compared to 1-, 3- and 6-month,12-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Herth, Principal Investigator — Thoraxklinik-Heidelberg gGmbH
Locations (1):
- Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided